CLINICAL TRIAL: NCT00781508
Title: Single Dose Sildenafil in Heart Failure Patients Improves 6-minute Walk Test by a Reduction in Left Ventricular Filling Pressure
Brief Title: Effects of Viagra on Heart Function in Patients With Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Robert Bahler, Cardiologist Professor of Medicine CWRU, MetroHealth Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MO1RR000080; Grant Number UL1 RR024989 (Other Grant/Funding Number: CWRU-CTSC); ULI RR024989 (Other Grant/Funding Number: NIH/NCRR CWRU-CTSC)
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Heart Failure; Left Ventricular Dysfunction
Keywords: heart failure, left sided; ventricular dysfunction; diastolic dysfunction; sildenafil
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left; Ventricular Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sildenafil (Experimental): Effect of oral administration of a single dose of sildenafil 50 mg on left ventricular filling pressures as evaluated 1 hr after sildenafil administration in patients with heart failure
  Interventions: Drug: sildenafil; Other: Placebo
- placebo (Placebo Comparator): Inactive placebo prepared to mimic the appearance of sildenafil.
  Interventions: Drug: sildenafil; Other: Placebo

INTERVENTIONS:
Drug: sildenafil — Changes in left ventricular filling pressure 1 hour after the administration of a single oral dose of sildenafil 50 mg.
  Other Names: Viagra
Other: Placebo — Changes in left ventricular filling pressure 1 hour after oral administration of placebo

SUMMARY:
Sildenafil (Viagra) is known to reduce pulmonary hypertension. Heart failure patients also have pulmonary hypertension and several recent reports have shown that sildenafil leads to an improvement in their exercise capacity. In these studies sildenafil caused a reduction in the pulmonary and systemic vascular resistances, improved pulmonary gas diffusion and perhaps increased cardiac output. It is uncertain if left ventricular filling pressures are reduced and whether there is improvement in left ventricular relaxation. The investigators hypothesize that in heart failure patients the improvement in exercise capacity associated with sildenafil is related to a significant reduction in left ventricular filling pressures. The investigators propose to study 20 patients with stable but moderately symptomatic heart failure. The study design is a randomized cross-over trial of the administration of a single dose of sildenafil 50 mg or a matching placebo. Exercise capacity will be determined before and after the oral administration of sildenafil 50 mg or placebo. Left ventricular filling pressures will be assessed by Doppler echocardiography and the serum level of B-type natriuretic peptide (BNP is known to increase with higher left ventricular filling pressures). After an initial echocardiogram and performing a 6 minute walk test, the patient will then be given either sildenafil or a matching placebo in a randomized double-blind fashion. One hr later a blood sample for serum BNP, the echocardiogram and the 6 minute walk test will be repeated.

DETAILED DESCRIPTION:
Sildenafil (Viagra) has been extensively studied in patients with idiopathic pulmonary hypertension. It reduces pulmonary vascular resistance, improves exercise capacity and is now an approved therapy for this condition. Heart failure (HF) patients also have pulmonary hypertension and several recent reports have shown that sildenafil leads to an improvement in their exercise capacity. In HF sildenafil causes a reduction in the pulmonary and systemic vascular resistances, improves pulmonary gas diffusion and perhaps increases cardiac output. It is uncertain if left ventricular filling pressures are reduced and whether there is improvement in left ventricular relaxation. We hypothesize that in HF patients the improvement in exercise capacity associated with sildenafil is related to a significant reduction in left ventricular filling pressures. We propose to study 10 patients with stable, symptomatic HF Class III. The study design is a randomized cross-over assignment of the administration of a single oral dose of sildenafil 50 mg or a matching placebo. Patients will be excluded if walking is impaired due to non-cardiac conditions or if they are taking nitrates. Exercise capacity will be determined before and 60 minutes after the oral administration of sildenafil 50 mg or placebo. The difference in the standardized 6 minute walk test (distance patient is able to walk over a 6 minute interval) will be used to assess exercise capacity. Left ventricular filling pressures will be assessed by Doppler echocardiography and the serum level of B-type natriuretic peptide (BNP). Evaluation of left ventricular relaxation will be determined by Doppler echocardiography techniques. Each patient will have a blood sample for BNP, an initial echocardiogram and perform a 6 minute walk test. They will then be given a single dose of either sildenafil or a matching placebo in a randomized double-blind fashion. The randomization was performed so that half of the group would receive the placebo on the initial test and sildenafil on the subsequent test and the other half would have the reverse sequence. One hr after the medication/placebo administration a blood sample for serum BNP, the echocardiogram and the 6 minute walk test will be repeated. After completion of the above protocol, the patient will return in 48 hrs and the protocol will be repeated with the predetermined assignment of either placebo or sildenafil.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Class III congestive heart failure and impaired left ventricular systolic function.
* A prior BNP level ≥ 200 pg/mL.
* Previously documented systolic pulmonary artery pressure >40 mmHg.
* Clinically stable for a minimum of 6 weeks.
* Able to give informed consent,

Exclusion Criteria:

* Unable to give informed consent.
* Currently taking nitrates.
* A HF exacerbation within the past 6 weeks.
* Co-morbid conditions that could limit their walking.
* Have a resting systolic blood pressure < 110 mmHg

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-12; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Bahler, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Heart Failure Clinic at MetroHealth Medical Center over a 12 month interval. Recruitment was slow due to the fact that many of the patients were already perscirbed nitrates and so were ineligible for the study.
Pre-assignment Details: More than 50 patients had to be excluded due to their already taking nitrates for their heart failure.
Groups:
- Sildenafil Then Placebo: Effect of sildenafil on left ventricular filling pressures in patients with heart failure
- Placebo Then Sildenafil: Effect of Sildenafil on left ventricular function
Period: Overall Study
Arm/Group | Sildenafil Then Placebo | Placebo Then Sildenafil
Started | 5 (First Intervention (1 day)", "Washout (48 hours)", "Second Intervention (1 day)) | 5 (First Intervention (1 day)", "Washout (48 hours)", "Second Intervention (1 day))
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sildenafil First Placebo Second: Effect of sildenafil on left ventricular filling pressures in patients with heart failure
- Placebo First Sildenafil Second: Effect of placebo on left ventricular filling pressures in patients with heart failure
- Total: Total of all reporting groups
Arm/Group | Sildenafil First Placebo Second | Placebo First Sildenafil Second | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (12) | 64 (12) | 64 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Reduction of the Left Ventricular Filling Pressure in Association With Administration of Sildenafil
Description: Left ventricular filling pressure was assessed by the ratio of the velocity of early mitral inflow (E) divided by the early tissue velocity (e). E/e
Time Frame: Left ventricular filling pressure was assessed 1 hr after oral administration of sildenafil
Population: All patients (10) that completed the protocol were analyzed.
Measure: Mean (Standard Deviation); unit: E/e' ratio
Groups:
- Sildenafil First Then Placebo: sildenafil 50 mg administered orally, placebo administered orally 48 hrs later
- Placebo First Then Sildenafil: placebo administered orally, then sildenafil orally 48 hrs later
Arm/Group | Sildenafil First Then Placebo | Placebo First Then Sildenafil
Number analyzed (Participants) | 5 | 5
E/e' ratio | 16.7 (6.9) | 16.4 (6.5)

2. Secondary Outcome: The Distance Walked During the 6-minute Walk Test 1 hr After the Oral Administration of Sildenafil 50 mg.
Description: A standardized course was used to determine the distance walked (meters) during a 6 min walk supervised by a nurse trained in performance of the test.
Time Frame: Measured 1 hr after oral administration of sildenafil 50 mg
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Sildenafil First Then Placebo: Sildenafil 50 mg orally, placebo orally 2 days later.
- Placebo First Then Sildenafil: placebo orally, then sildenafil 50 mg orally 2 days later.
Arm/Group | Sildenafil First Then Placebo | Placebo First Then Sildenafil
Number analyzed (Participants) | 5 | 5
meters | 210 (34) | 219 (40)

ADVERSE EVENTS:
Time Frame: The study took place over a 1 year interval
Description: Patients were observered for any side effects or adverse reactions for 2 hrs following the administration of either sildenafil or placebo.
Groups:
- Sildenafil First Then Placebo: Effect of sildenafil first on left ventricular filling pressures, then effect of placebo on left ventricular filling pressure
- Placebo First Then Sildenafil: Effect of placebo on left ventricular filing pressures, then effect of sildenafil on left ventricular filling pressure.
Arm/Group | Sildenafil First Then Placebo | Placebo First Then Sildenafil
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
The study was limited by the small number of participants. Additionally, the inclusion criterion of a systolic pulmonary artery pressure of > 40 mmHg was no longer present in the majority of patients at the time they presented for study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No